CLINICAL TRIAL: NCT05495633
Title: SteamOne - Prospective Database for Rezum Water Vapor Therapy of the Prostate
Acronym: SteamOne
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-00544; bb21Ebbing
Record Dates: First submitted 2022-07-18; First posted 2022-08-10 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Benign Prostate Obstruction (BPO)
Keywords: Lower Urinary Tract Symptoms (LUTS); Rezum water vapor therapy; prostate
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — Patient Reported Outcome Measures; Amyloid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Collection and evaluation of clinical (CROMs) and patient-reported outcomes (PROMs) — The study uses a web-based German-language database (electronic data capture system, EDCS) called "REDCap" that provides both clinical reported outcome measures (CROMs) and patient-reported outcome measures (PROMs). PROMs are investigated by validated questionnaires: IPSS/QoL, ICIQ-MLUTS, MSHQ, ICIQ-MLUTSsex, QoR-15GE, PROMIS Global Health 10, ICIQ-S, NRS, and by home urine flow measurement (initially iUFlow, since October 2025 EmanoFlow ) as well as by self-designed questionnaires to assess patients´ preferences and expectations for Rezum and for surgical therapy of the prostate, satisfaction with the Rezum therapy, side effects of the Rezum therapy, (re)medication to treat BPO and LUTS, and reoperations after Rezum therapy.
Other: Analysis of uroflowmetry data by EmanoFlow Mobile Application (App) and Emano Clinic Portal — If patients have a smartphone with app function (Android or Apple), they will be provided with an FDA-registered home uroflowmetry mobile App (called EmanoFlow from Emano Metrics, USA) at study entry. This AI-based mobile application should enable patients to measure their urine flow conveniently from home and thus be independent of the medical consultation. EmanoFlow is marketed by Emano Metrics Inc., a Delaware C Corporation with its principal place of business at 132 East Broadway Suite 700, Eugene, OR, 97401, USA. Every time a patient is using the mobile App urine flow measurement data will be sent to the home uroflowmetry database (Emano Flow Clinic Portal).

SUMMARY:
This study is to assess the clinical data of Rezum (water vapor therapy) in patients with BPO (benign prostate obstruction) and male LUTS (lower urinary tract symptoms) in terms of efficacy, durability and safety in a large, prospective, multi-center cohort consisting of 1000 "real-life" patients with a follow-up of 5 years.

DETAILED DESCRIPTION:
Prostate water vapor therapy (Rezum) is an approved treatment procedure for the management of lower urinary tract symptoms in men caused by benign prostatic obstruction (BPO). Rezum is performed transurethrally by steam injections into the central or transition zone of the enlarged prostate. The 103°C hot steam is generated by a generator and injected into the prostate tissue via a disposable handpiece with a retractable needle. Approximately 1 injection is required per 10 ml of prostate tissue to achieve desobstruction. The single injection takes only 9 seconds. The thermal energy contained in the water vapor is able to develop evenly and freely in the intercellular space of the prostate by convection. This represents a unique technique in surgical desobstruction of the prostate. The steam condenses and releases the stored heat energy to the cell membranes, which then denature. As a result, the prostate tissue shrinks by about 30% in the first three months after the Rezum treatment. The shrinkage process therefore does not take place immediately, but with a time delay. The minimally invasive nature of the procedure results from the short surgical time, the potential of Rezum to preserve sexual function (both ejaculation and erection), and the possibility of performing Rezum even under local anesthesia or analgesia. Data on efficacy, durability of efficacy, safety/complications, and indication groups are still limited. "Real life" data are important to determine the role of Rezum water vapor therapy in the treatment of BPO and male LUTS. The aim of this study is to prospectively enroll and follow Rezum patients in a multicenter, German-language, web-based database. Patient-reported outcome measures (PROMs) and clinical-reported outcome measures/data (CROMs) on various subgroups of patients treated with Rezum as a routine clinical treatment option for BPO-related male LUTS will be recorded in terms of procedure efficacy, functional outcomes (e.g. sexual function) and surgical safety. Further aspects of interest are recovery from the procedure, patients' expectations towards Rezum treatment, patients' satisfaction with Rezum treatment, and impact of Rezum on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* All male patients who are treated with Rezum due to prostate obstruction and LUTS in the participating study centers can be included if certain inclusion criteria are met and some exclusion criteria are not present.
* The indication to perform Rezum needs to be made independently from the study. The decision for Rezum treatment is the responsibility of each individual practitioner and patient.
* Age ≥ 18 years
* Operated or supervision of surgery by a certified urologist
* Subgroups of special interest are e.g. catheter-dependent patients, patients with oral anticoagulation, patients with preoperative urodynamic pressure-flow investigation (not older than 6 months) or patients with prostates bigger than 80 ml

Exclusion Criteria:

* Missing informed consent
* Lack of ability to answer questionnaires due to laguage problems or mental incapacity (e.g. in dementia, mental disability)
* Patient does not have a personal email address available and the survey cannot be completed via a relative's email address and the patient is not willing to complete the survey on the tablet at the clinic
* Known or suspected neurogenic bladder dysfunction in e.g. Parkinson's disease, multiple sclerosis or other neurological diseases with possible effects on bladder function
* History of malignant bladder tumor in the last two years (including CIS) or currently present malignant bladder tumor at time of Rezum treatment (including CIS)
* Previous operation(s) on the prostate, except prostate biopsy, if this was performed more than 4 weeks ago at time of Rezum treatment
* Previous operation(s) on the bladder neck
* Presence of bladder neck stenosis requiring treatment at time of Rezum treatment
* Planned combination of Rezum treatment concurrently with another urologic (*) or non-urologic procedure

(*) also the combination with a planned transurethral procedure is not allowed except for bladder stone removal

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are treated with Rezum - water vapor therapy of the prostate due to benign prostate obstruction (BPO) or male lower urinary tract symptoms (LUTS) as part of routine clinical practice. Patients will be recruited within the participating study hospitals as part of regular patient care after an indication for Rezum treatment has been made independent of the study.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-12-16 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Change in International Prostate Symptom Score/ Quality of Life (IPSS/ QoL) | At baseline, 6 weeks, 3 months, 6 months, 12 months and annually until the 5th follow-up year after treatment with Rezum
  The IPSS is an eight-item validated questionnaire, consisting of seven symptom questions and one QoL question. The IPSS score is categorised as 'asymptomatic' (0 points), 'mildly symptomatic' (1-7 points), 'moderately symptomatic' (8-19 points), and 'severely symptomatic' (20-35 points).

SECONDARY OUTCOMES:
Change of maximum urinary flow rate (Qmax) measured by uroflowmetry | At baseline, 2 weeks, 6 weeks, 3 months, 6 months, 12 months and annually until the 5th follow-up year after treatment with Rezum
  Self-measured by patients at home using the iUFlow device (Kesem Health)
Change of International Consultation on Incontinence Questionnaire for male lower urinary tract symptoms (ICIQ-MLUTS) | At baseline, 6 weeks, 3 months, 6 months, 12 months and annually until the 5th follow-up year after treatment with Rezum
  The ICIQ-MLUTS is a widely used and validated patient-completed questionnaire including incontinence questions and bother for each symptom. It contains thirteen items (including incontinence questions and bother for each symptom), with subscales for nocturia and overactive bladder (OAB).
Change of Male Sexual Health Questionnaire (MSHQ) | At baseline, 6 weeks, 3 months, 6 months, 12 months and then annually until the 5th follow-up year after treatment with Rezum
  The MSHQ long form includes 3 domains: Erection scale (3 items), Ejaculation scale (7 items), Sexual satisfaction scale (6 items) (additional 2 items measuring bothersome linked to erection and ejaculation). Additional Items (Sexual Activity and Desire) are not to be collected.
Change of International Consultation on Incontinence Questionnaire Male Sexual Matters Associated with Lower Urinary Tract Symptoms Module (ICIQ-MLUTSsex) | At baseline, 6 weeks, 3 months, 6 months, 12 months and then annually until the 5th follow-up year after treatment with Rezum
  The ICIQ-MLUTSsex is a patient-completed questionnaire for detailed evaluation of male sexual matters associated with their lower urinary tract symptoms and impact on quality of life (QoL). It is composed of 4 sections (erection, ejaculation, pain/discomfort during ejaculation, impact of urinary symptoms).
Patient's postoperative recovery by QoR-15 | At baseline, at the first postoperative day and 2 weeks after treatment with Rezum
  Investigation of type of anesthesia (general anesthesia, spinal anesthesia, local anesthesia, analgosedation) incl. reason for type of anesthesia and postoperative recovery using the validated German version of the Quality-of-Recovery-Score (QoR-15GE).
Change in PROMIS Global Health 10 questionnaire | At baseline, 2 weeks, 6 weeks, 3 months, 6 months, 12 months and then annually until the 5th follow-up year after treatment with Rezum
  Changes in Quality of Life associated with Rezum treatment using the PROMIS Global Health 10 questionnaire. It is a measure of overall health-related quality of life. The questionnaire consists of a combination of 10 questions that assess both the physical and mental health status of adult patients independent of their individual medical situation. The items are measured using a five-point response matrix that includes physical function, fatigue, pain, emotional distress and social health.
Change in ICIQ-S (International Consultation on Incontinence - Satisfaction) | At 2 weeks, 6 weeks, 3 months, 6 months, 12 months and annually after treatment with Rezum
  The ICIQ-S (International Consultation on Incontinence - Satisfaction) will be used to evaluate patient satisfaction after urological surgery. Question items consist of: outcome success, comparison of symptoms, return to "normal life", same situation, same choice, recommend, current symptoms, preparation for surgery, satisfaction of explanation, pain after surgery, satisfaction of pain relief, current pain, complications/side effects, result of surgery and satisfaction with surgery.
Numeric pain Rating Scale (NRS) | At the first postoperative day
  Investigation of patients' perception of pain during Rezum procedure in case of local anesthesia and/or analgosedation and after Rezum treatment using NRS. The NRS has the following scale: from 0 - 10 (no pain - worst pain imaginable).
Rezum side effects and Pain medication | At baseline, 2 weeks, 6 weeks and 3 months
  This questionnaire is self-designed. Typical side effects must be seen and investigated independently of treatment complications in order to provide patients with the best possible advice and information. The need for pain medication will be evaluated in a time context as well.
Patients' preferences and expectations of Rezum Treatment | At baseline, 3 months, 6 months, 12 months and then annually until the 5th follow-up year after treatment with Rezum
  This self-designed questionnaire considers measurement tools related to BPO/male LUTS treatment and aims to investigate patients' motivations, expectations and preferences for surgical desobstruction of the prostate due to BPO in general but also in particular concerning the Rezum treatment. This will attempt to better understand patient attitudes in order to improve future counseling of patients regarding minimally invasive procedures for the treatment of BPO-related male LUTS.
Questionnaire: BPO (BPH)/LUTS medication | At 2 weeks, 6 weeks, 3 months, 6 months, 12 months and then annually until the 5th follow-up year after treatment with Rezum
  This self-designed questionnaire aims to evaluate the need for BPO (BPH)/LUTS medication.
Questionnaire: Reoperation | At 3 months, 6 months, 12 months and then annually until the 5th follow-up year after treatment with Rezum
  This self-designed questionnaire aims to evaluate the need for urological reoperation.
Questionnaire: Bladder catheter | At 3 months, 6 months, 12 months and then annually until the 5th follow-up year after treatment with Rezum
  This self-designed questionnaire aims to evaluate the need for bladder catheterization.
Number of steam injections and injection points during Rezum treatment | At Baseline (on day of treatment with Rezum)
  Investigation of the influence of the number of steam injections and Injection points on outcome parameters, micturition parameters, sexual function, prostate size, side effects and complications.
Retreatment rate | Up to 5 years after treatment with Rezum
  Number of retreatments (medical (drugs), bladder catheter and surgical) after Rezum treatment.
Surgical safety by classification of intraoperative adverse events (ClassIntra®) | On day of treatment with Rezum
  The classification defines intraoperative adverse events as any surgery or anesthesia-related deviation from the ideal intraoperative course occurring between begin of anesthesia and end of anesthesia.
  Surgical safety is investigated by analyzing intraoperative complications classified by ClassIntra (from Grade 0: No deviation from the ideal intraoperative course to Grade 5: Any deviation from the ideal intraoperative course with intraoperative death of the patient).
30-days postoperative complications by the Clavien-Dindo classification | Within 30-days after treatment with Rezum
  The classification defines postoperative adverse events occurring after the patient has left the recovery room until 30 days after surgery (from Grade I: Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological intervention to Grade V: Death of a patient).
Antimicrobial prophylaxis | Within the first 30 days after treatment with Rezum
  Investigation of the effectiveness of the chosen antimicrobial prophylaxis by analyzing the rate of postoperative symptomatic urinary tract infections (UTI) within the first 30 days after surgery as part of the Clavien-Dindo classification. Definition of symptomatic UTI is based on clinical diagnosis supported by measured bacteriuria of ≥105 cfu/ml treated with antimicrobial agents.
Post voiding residual volume (PVR) measured by ultrasound | Baseline and up to 5 years after treatment with Rezum
  Change of post voiding residual volume (PVR) measured by ultrasound is a simple test that can raise or lower the suspicion of bladder outlet obstruction (BOO).
Change of prostate size | Baseline and up to 5 years after treatment with Rezum
  Measured by ultrasound or magnetic resonance imaging (MRI).
Change in bladder outlet obstruction index (BOOI) | Max. 6 months before Rezum and/or 3-6 months after Rezum treatment
  BOOI is represented by the equation: BOOI = Pdet @ Qmax - 2 x Qmax (Pdet = detrusor pressure; Qmax = maximum flow rate). BOOI > 40 = obstructed; BOOI 20-40 = equivocal; and BOOI < 20 = unobstructed.
Change in bladder contractility index (BCI) | Max. 6 months before Rezum and/or 3-6 months after Rezum treatment
  The BCI is represented by the following formula: BCI = Pdet @ Qmax + 5 x Qmax. Using this formula, contractility can be divided into strong > 150, normal 100-150, and weak < 100.
Change in International Prostate Symptom Score (IPSS) for detrusor (bladder muscle) overactivity (DO) | Max. 6 months before Rezum and/or 3-6 months after Rezum treatment
  Urodynamic analysis of detrusor overactivity (DO) during storage phase and correlation of pre- and postoperative DO with PROMs (IPSS). The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
MRI (magnetic resonance imaging) data | Max. 12 months before Rezum and up to 5 years after treatment with Rezum
  MRI data not older than 12 months at time of Rezum treatment and MRI data in the follow-up period of 5 years are investigated in terms of prostate size, ablative lesions (lesions caused by Rezum) and PI-RADS (prostate imaging-reporting and data system) lesions.
Prostate cancer (PCa) detected by positive prostate biopsy | Max 12 months and up to 5 years after treatment with Rezum
  The proportion of patients who receive Rezum treatment with a history of prostate cancer or who develop histologically confirmed prostate cancer during the post-treatment course.
Doctors' preferences, motivations and reasons to use Rezum | Before treatment with Rezum
  Investigation of doctors' reasons for preference/choice of using Rezum in a patient using a self-designed questionnaire.
Change in ICIQ-Lower Urinary Tract Symptoms Quality of Life (ICIQ-MLUTS) score for detrusor (bladder muscle) overactivity (DO) | Max. 6 months before Rezum and/or 3-6 months after Rezum treatment
  Urodynamic analysis of detrusor overactivity (DO) during storage phase and correlation of pre- and postoperative DO with PROMs (ICIQ-MLUTS). The ICIQ-MLUTS is a questionnaire for evaluating male lower urinary tract symptoms and impact on quality of life (QoL). 1-84 overall score with greater values indicating increased symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Ebbing, PD Dr. med., Principal Investigator — University Hospital Basel, Department of Urology
Locations (19):
- Universitätsklinikum Graz, Graz, Austria
- Germany (10):
  - Alexianer St. Hedwig-Krankenhaus, Berlin
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Hamburg-Eppendorf (UKE),, Hamburg
  - Asklepios Westklinikum Hamburg GmbH, Hamburg
  - Urologische Gemeinschaftspraxis Prüner Gang, Kiel
  - Krankenhaus Maria Hilf - Alexianer Krefeld, Krefeld
  - Klinikum Nürnberg, Nuremberg
  - Krankenhaus Reinbek St. Adolf Stift, Reinbek
  - Kliniken Sindelfingen, Sindelfingen
  - Diakonie-Klinikum Stuttgart Diakonissenkrankenhaus und Paulinen gGmbH, Stuttgart
- Switzerland (8):
  - Kantonsspital Aarau, Aarau, Aarau
  - Hirslanden Klinik St. Anna, Lucerne, Canton of Lucerne
  - University Hospital Basel, Department of Urology, Basel
  - Inselspital Bern, Bern
  - Kantonsspital Luzern, Lucerne
  - Uroviva AG, Rothrist
  - Kantonsspital St. Gallen, Sankt Gallen
  - Universitätsspital Zürich, Zurich

REFERENCES:
- See also: SteamOne Homepage (German Language) — https://www.unispital-basel.ch/urologie/forschung-urologie/steamone

DOCUMENTS (2):
  • Study Protocol (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/33/NCT05495633/Prot_003.pdf
  • Statistical Analysis Plan (2021-09-29): https://cdn.clinicaltrials.gov/large-docs/33/NCT05495633/SAP_001.pdf